CLINICAL TRIAL: NCT03520179
Title: Improving Standards of Care and Translational Research in Spinal Muscular Atrophy (SMA)
Acronym: SMA-REACH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 11DN15
Record Dates: First submitted 2018-01-30; First posted 2018-05-09 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SMA TYPE 1: genetically confirmed SMA
- SMA TYPE 2: genetically confirmed SMA
- SMA TYPE 3: genetically confirmed SMA, Ambulant and non-ambulant

SUMMARY:
The SMA REACH UK Network is a national and international partnership between doctors and therapists involved in the care of children and adults with Spinal Muscular Atrophy. This network is supported by Biogen and SMA UK.

DETAILED DESCRIPTION:
The investigators aim is to establish a Spinal Muscular Atrophy (SMA) National Platform to improve UK standards of care, manage national and International clinical trials and facilitate translational research for this common neuromuscular disease.

To achieve this purpose investigators will start to systematically collect longitudinal validated outcome measures for SMA children followed at GOSH, the largest cohort followed in UK, and pilot and update novel outcome measures. This will be done ensuring that data collected are not only clinically meaningful but also robust for subsequent use in clinical trials.

In collaboration with the MRC Neuromuscular Centre in London and Newcastle, investigators will link the existing registries and the longitudinal data collection of outcome measures and develop a hub and bespoke platform model linking the other paediatric UK centres involved in the clinical management of SMA patients. This UK SMA Platform (SMA REACH UK) will be a unique infrastructure containing the largest comprehensive longitudinal series of SMA patient data in the UK; the data collected will be agreed between the relevant other UK centres stakeholders and will take into consideration other international initiatives with historical success in SMA treatment and research.

Ongoing analysis including modern psychometric techniques will ensure that the functional data collected in the UK SMA population meets the high statistical standards required for the data to inform natural history studies and be usable as an outcome measure for clinical trials.

In addition SMA REACH UK is in the position to be involved in an international initiative called ISMAC (International SMA Consortium) with two prestigious Networks: the PNCRN in the United States (Principal Investigator Richard Finkel) and the Italian SMA Network (Principle Investigator Eugenio Mercuri). The Consortium has been contacted by the Biotechnology Company; Biogen with strong interest in collecting anonymised natural history data on the entire spectrum of SMA severity from routine clinical visits. The main data to be collected, including medical information and physiotherapy assessments, were agreed across the three Networks and will be slightly more extended than the current dataset collected at each Centre. The data collected with the new dataset will be collated on a separate IT platform which will contain anonymised clinical and physiotherapy data from patients who have consented to take part, and will be accessible to Biogen and can be shared with third parties (pharmaceuticals, academic and government institutions) in a strictly anonymised form. The ownership of the data will remain with the PIs at each centre.

ELIGIBILITY:
Inclusion Criteria:

* It will be genetically confirmed SMA

Exclusion Criteria:

* Involvement in clinical trials is not an exclusion criterion nor having had surgical procedures. Patients who are participating in clinical trials with novel treatments will also be included in the database although the data from this subgroup won't be analysed in the natural history study, nor shared with pharmaceutical companies and other third parties as part of the ISMAC collaboration.

Ages: 0 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with genetically confirmed SMA types 0, I, II and III (ambulant and non-ambulant) followed at each open and recruiting neuromuscular centre.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2013-12-17 (Actual); Primary Completion 2023-08-12 (Estimated); Study Completion 2023-08-12 (Estimated)

PRIMARY OUTCOMES:
Physiotherapy assessment using The Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND) | 1 year
  This is a scale used for the assessment of movement and function of very weak infants with SMA type 1. It consists of 16 items of motor function graded 0-4 with a maximum achievable score of 64.
Physiotherapy assessment using the Test of Infant Motor Performance Screening Items (TIMPSI) | 1 year
  This scale assesses motor performance in infants born pre-term to 4 months of age. It consists of 29 items, with 3 item sets (screening, easy and hard sets).

SECONDARY OUTCOMES:
Patient´s perception about the condition, interventions performed and Standards of Care assessed by patient interviews | 1 year
  The patients will be selected depending on availability and willingness to participate.The interviews will be performed at the most convenient time for the patient. They will be done either face to face, through a phone call or videoconference.
Patients perception about the condition, interventions performed and Standards of Care assessed using the Paediatric Outcomes Data Collection Instrument (PODCI) | 1 year
  This is a questionnaire which assesses overall health, pain and ability to participate in activities of daily living. It can be scored relating to eight scales - upper extremity and physical function, transfers and basic mobility, sports/physical functioning, pain/comfort, treatment expectations, happiness, satisfaction with symptoms, global functioning.
Patients perception about the condition, interventions performed and Standards of Care assessed using the Egan Klassifikation Scale (EK2) | 1 year
  This is a questionnaire to be used for non-ambulant patients and consists of a series of 17 questions reporting on physical function including ability to transfer, cough, swallowing, fatigue and arm function.

CONTACTS AND LOCATIONS:
Locations (1):
- Dubowitz Neuromuscular Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No